CLINICAL TRIAL: NCT04148625
Title: Subxyphoid Epicardial/Endocardial Hybrid Atrial Fibrillation Ablation and Left Atrial Appendage (LAA) Exclusion Approach for Patients With Persistent and Longstanding Persistent Atrial Fibrillation Registry
Brief Title: Subxyphoid Hybrid MAZE Registry for Patients With Persistent Atrial Fibrillation
Acronym: SubXMAZE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of California, San Francisco (Other)
Collaborators: Vanderbilt University Medical Center (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 19-29483
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: hybrid, LAA ligation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- atrial fibrillation, persistent: Subjects with documented symptomatic persistent or longstanding persistent AF (> than 3 months and < 3 years continuous AF duration) who has failed a previous PVI catheter ablation procedure and/or needs LAA exclusion; and catheter ablation or minimally surgical approach is planned.

SUMMARY:
Minimally invasive surgical procedures have been advocated as an alternative to catheter ablation for the treatment of persistent atrial fibrillation. Initial results have been promising in maintaining sinus rhythm compared to catheter ablation, but are associated with a considerably greater number of procedural-related adverse events compared to catheter ablation. This study investigates the safety and feasibility of a new subxyphoid epicardial/endocardial hybrid atrial fibrillation ablation and LAA exclusion approach for patients with persistent and longstanding persistent atrial fibrillation.

DETAILED DESCRIPTION:
The study will assess the ability of a subxyphoid and percutaneous hybrid epicardial/endocardial ablation approach consisting of pulmonary vein isolation (PVI), LAA exclusion, isolation of the left atrial (LA) posterior wall and cavotricuspid isthmus (CTI) line (Hybrid Sub-X MAZE) to (1) demonstrate that the hybrid procedure does not result in an unacceptable risk of serious adverse events (SAEs) in persistent or longstanding persistent atrial fibrillation (AF) subjects for whom an ablation procedure is planned; and (2) assess freedom from episodes of persistent AF > 30 seconds duration during the observation period through 12 months post PVI.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for the study:

1. Age ≥ 18 years and ≤ 80 years at time of screening.
2. Documented diagnosis of symptomatic persistent or persistent longstanding non-valvular atrial fibrillation

   * Persistent AF is defined as atrial fibrillation sustained for ≥ 7 days and ≤ 1 year;
   * Longstanding persistent AF is defined as continuous atrial fibrillation > 1 year duration;
   * Non-valvular atrial fibrillation is defined as cases without a mechanical heart valve requiring anticoagulation or without moderate to severe mitral stenosis.

   Note: Persistent AF and Longstanding Persistent AF must be documented as follows:

   Persistent AF:
   * Physician's note indicating that patient has experienced symptomatic continuous AF that is sustained ≥ 7 days duration and < 1 year and clinical history of non-paroxysmal AF < 3 years; and
   * A ≥7-day continuous rhythm monitoring (e.g., Zio patch, implantable loop recorder (ILR), pacemaker) which documents 90% AF burden over at least 7 consecutive days or alternatively, two electrocardiograms from any form of rhythm monitoring (e.g. 12-lead ECG, Holter, event monitor) documenting continuous AF, with electrocardiograms taken at least 7 days apart, for subjects with sustained AF ≥ 7 days, as confirmed by the ECG Core Laboratory, obtained within 90 days prior to randomization.

   Longstanding Persistent AF:
   * Physician's note indicating that patient has experienced symptomatic continuous AF that is sustained > 1 year duration and clinical history of non-paroxysmal AF < 3 years; and
   * A ≥7-day continuous rhythm monitoring (e.g., Zio patch, ILR, pacemaker) which documents 90% AF burden over at least 7 consecutive days or alternatively, 24 hour continuous rhythm monitoring (e.g. holter, event monitor) obtained within 90 days prior to the index procedure showing continuous AF, as confirmed by the ECG Core Laboratory. Note: The performance of a successful cardioversion (sinus rhythm ≥30 seconds) within 12 months of an ablation procedure with documented early recurrence of AF within 30 days should not alter the classification of AF as Longstanding Persistent.)
3. Failed previous catheter PVI ablation
4. Life expectancy ≥ 1 year;
5. Willing and able to return to and comply with scheduled follow-up visits and tests; and
6. Willing and able to provide written informed consent

Exclusion Criteria:

Exclusion Criteria: Subjects will be excluded if he / she meets any of the following:

1. Prior procedure involving opening of the pericardium or entering the pericardial space (e.g., coronary artery bypass graft (CABG), heart transplantation, valve surgery) where adhesions are suspected;
2. Measured LA diameter > 6.5 cm;
3. Documented embolic stroke, Transient ischemic attack (TIA) or suspected neurologic event within 3 months prior to the planned intervention;
4. Currently exhibits New York Heart Association (NYHA) Class IV heart failure symptoms;
5. Documented history of right heart failure specifically when right ventricle exceeds the left ventricular size;
6. Documented history of myocardial infarction (MI) within 3 months prior to the planned study intervention;
7. Documented history of unstable angina within 3 months prior to the planned study intervention;
8. Recent documented history of cardiogenic shock, hemodynamic instability or any medical condition in which intra-aortic balloon pump (IABP) therapy is clinically indicated;
9. Documented symptomatic carotid disease, defined as > 70% stenosis or > 50% stenosis with symptoms;
10. Diagnosed active local or systemic infection, septicemia or fever of unknown origin at time of baseline screening;
11. Chronic renal insufficiency defined as estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 within 3 months prior to study treatment;
12. End Stage Renal Disease (ESRD) or documented history of renal replacement / dialysis;
13. Current documented history of clinically significant liver disease which predisposes the subject to significant bleeding risk (clinically defined by the treating physician);
14. Any history or thoracic radiation with the exception of localized radiation treatment for breast cancer;
15. Current documented use of long-term treatment with corticoid steroids, not including use of inhaled steroids for respiratory diseases;
16. Active pericarditis;
17. Active endocarditis;
18. Any documented history or autoimmune disease associated with pericarditis;
19. Evidence of Pectus Excavatum (documented and clinically defined by the treating physician);
20. Untreated severe scoliosis (documented and clinically defined by treating physician);
21. Thrombocytopenia (platelet count < 100 x 109/L) based on most recent pre-procedure assessment within 30 days prior to planned intervention;
22. Anemia with hemoglobin concentration of <8 g/dL based on most recent pre-procedure assessment (within 30 days prior to planned intervention);
23. Left Ventricular Ejection Fraction (LVEF) < 30% within 30 days prior to planned intervention;
24. Known acquired or inherited propensity for forming blood clots (e.g., malignancy, Factor V leiden mutation) established by prior objective testing;
25. Documented presence of implanted congenital defect closure devices, (e.g., atrial septal device (ASD), patent foramen vale (PFO) or ventricular septal device (VSD) device);
26. Previously attempted occlusion of the LAA (by any surgical or percutaneous method);
27. Inability, unwillingness or contraindication to undergo TEE imaging;
28. Body Mass Index (BMI) > 40;
29. Evidence of active Graves disease;
30. Current untreated hypothyroidism;
31. Any contraindication to suture, endovascular device, or other minimally invasive techniques including percutaneous, transseptal, and/or sub-xiphoid access.
32. Subject is pregnant or plans / desires to get pregnant within next 12 months;
33. Current enrollment in an investigation or study of an investigational device or investigational drug that would interfere with this study and the required follow up;
34. Mental impairment or other psychiatric conditions which may not allow patient to understand the nature, significance and scope of the study;
35. Any other criteria, medical illness or comorbidity which would make the subject unsuitable to participate in this study as determined by the clinical site Primary Investigator; Additional Exclusion Criteria: Based on Screening / Pre-procedure Imaging

Subjects will also be excluded if they meet any of the following:

1. Based on screening computed tomography angiography (CTA) performed prior to study intervention:

   * LAA Morphology: Superior-posterior oriented LAA (i.e. superior C shape), that has:

     1. LAA LARIAT-approach width ≥ 40 mm; or
     2. LAA distal apex extending posterior to the ostium of the LAA.
   * LAA positioned behind the pulmonary artery; or
   * All other LAA morphology: LAA LARIAT approach width > 45 mm.
2. Based on a peri-procedural imaging (TEE at time of hybrid sub-X MAZE procedure. or catheter ablation):

   * Intracardiac thrombus; or
   * Significant mitral valve stenosis (i.e., mitral valve (MV) stenosis < 1.5cm2)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with documented symptomatic persistent or longstanding persistent AF (> than 3 months and < 3 years continuous AF duration) who has failed a previous PVI catheter ablation procedure and/or needs LAA exclusion; and catheter ablation or minimally surgical approach is planned.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-09-14 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from episodes of AF > 30 seconds | 12 months
  * No evidence of any episode of AF/AT/AFL > 30 seconds duration, as documented by 24 hour holter monitoring at any time following the 90-day blanking period post index PVI at 6 and 12 months; and/or if patient has symptoms of palpitations.
  * No additional catheter ablation procedures post index PVI (aside from ablation for right-sided AFL)
  * No requirement for new Class I or III anti-arrhythmic drug (AAD) prescribed to treat atrial fibrillation following day 120 (90 day blanking period + 30 day window).
The incidence of adjudicated significant device- or procedure-related SAEs • Pericardial effusions requiring surgical intervention occurring within 30 days after the hybrid sub-X MAZE procedure. | 30 days after hybrid procedure• Pneumothorax requiring surgical treatment • Vascular Injury requiring surgical treatment
  • Serious injury to cardiac/ related structure requiring surgical intervention• Bleeding• Pericarditis requiring surgical treatment• Hemothorax requiring surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Lee, MD, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Badhwar N, Al-Dosari G, Dukes J, Lee RJ. Subxiphoid Hybrid Approach for Epicardial/Endocardial Ablation and LAA Exclusion in Patients with Persistent and Longstanding Atrial Fibrillation. J Atr Fibrillation. 2018 Jun 30;11(1):2014. doi: 10.4022/jafib.2014. eCollection 2018 Jun-Jul. PMID 30455837
- [Result] Sanchez JM, Al-Dosari G, Chu S, Beygui R, Deuse T, Badhwar N, Lee RJ. Hybrid and surgical procedures for the treatment of persistent and longstanding persistent atrial fibrillation. Expert Rev Cardiovasc Ther. 2018 Feb;16(2):91-97. doi: 10.1080/14779072.2018.1425140. Epub 2018 Jan 12. PMID 29327638